CLINICAL TRIAL: NCT07406672
Title: Evaluation of Differences Between Joint Localizations Determined by Physical Examination and Ultrasound-Confirmed Joint Positions of the Knee, Elbow, Ankle and Wrist
Brief Title: Comparison of Clinical Joint Localization and Ultrasound-Confirmed Joint Positioning
Status: Not yet recruiting | Type: Observational
Sponsor: Bursa City Hospital (Other Government)
Responsible Party: Principal Investigator, Taner Dandinoğlu, Principal Investigator, Bursa City Hospital
Other Study IDs: 2026-PMR-3
Record Dates: First submitted 2026-02-06; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Musculoskeletal System; Physical Examination
Keywords: Ultrasonography; Musculoskeletal Ultrasound; Clinical Anatomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Physician Participants: Volunteer physicians working as residents or specialists in Physical Medicine and Rehabilitation or Orthopedics and Traumatology who undergo clinical joint localization assessment and ultrasound confirmation.
  Interventions: Other: Observational Assessment

INTERVENTIONS:
Other: Observational Assessment — No therapeutic or diagnostic intervention is applied. Participants undergo an observational assessment consisting of physical examination-based joint localization followed by ultrasound confirmation for measurement and comparison purposes only.

SUMMARY:
This prospective, cross-sectional observational study aims to evaluate the differences between joint localizations determined by physicians based on physical examination and joint positions confirmed by musculoskeletal ultrasound. Knee, elbow, ankle, and wrist joints will be assessed in volunteer physicians working in Physical Medicine and Rehabilitation and Orthopedics and Traumatology.

For each joint, participants will identify the joint space based on physical examination and the marked locations will be compared with ultrasound-confirmed joint positions. The distance between clinically determined and ultrasound-confirmed locations will be measured in millimeters. The study seeks to provide objective data on the accuracy of clinical joint localization and to support educational approaches in clinical anatomy and musculoskeletal examination training.

DETAILED DESCRIPTION:
This study is designed as a prospective, cross-sectional, observational comparison of clinical joint localization and ultrasound-confirmed joint positioning. The study will be conducted at Bursa City Hospital and will include volunteer physicians working as residents or specialists in Physical Medicine and Rehabilitation or Orthopedics and Traumatology.

Participants will be asked to localize the joint space of the knee (tibiofemoral), elbow (humeroulnar), ankle (tibiotalar), and wrist (radiocarpal) based on physical examination in standardized positions. Clinically determined joint locations will be marked on the skin using a removable marker.

Following clinical marking, musculoskeletal ultrasound examinations will be performed by an experienced investigator using a high-frequency linear transducer. Ultrasound-confirmed joint positions will be identified according to standardized scanning protocols. The investigator performing the ultrasound assessment will be blinded to the participant's specialty and level of experience.

The primary outcome measure will be the distance, measured in millimeters, between the clinically marked joint location and the ultrasound-confirmed joint position. Secondary analyses will evaluate differences in localization accuracy among different joints and between physicians with different levels of clinical experience.

The study involves no therapeutic or diagnostic intervention and poses minimal risk to participants. All data will be collected anonymously and analyzed at the group level. The results are expected to contribute to a better understanding of the limitations of physical examination-based joint localization and to inform educational strategies incorporating ultrasound in clinical anatomy training.

ELIGIBILITY:
Inclusion Criteria:

* Physicians working as residents or specialists in Physical Medicine and Rehabilitation or Orthopedics and Traumatology
* Age 18 years or older
* Voluntary participation with written informed consent
* Ability to perform physical examination-based joint localization

Exclusion Criteria:

* Refusal to participate or provide written informed consent
* Any condition preventing completion of physical examination procedures
* Non-compliance with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult physician volunteers recruited from a tertiary care hospital. Participants are licensed medical doctors who participate as reference subjects for joint localization. Each participant is asked to indicate the anatomical location of selected joints (knee, elbow, ankle, and wrist), which is subsequently assessed by physical examination and confirmed using ultrasound imaging within the scope of this observational study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Distance Between Clinically Determined and Ultrasound-Confirmed Joint Localization | Single assessment session
  The distance, measured in millimeters, between the joint location identified by physical examination and the joint position confirmed by musculoskeletal ultrasound.

SECONDARY OUTCOMES:
Joint-Specific Differences in Localization Accuracy | Single assessment session.
  Comparison of distance differences between clinically determined and ultrasound-confirmed joint localization across different joints (knee, elbow, ankle, and wrist).
Effect of Physician Experience on Joint Localization Accuracy | Single assessment session
  Comparison of distance differences between clinically determined and ultrasound-confirmed joint localization according to physician experience level (resident versus specialist).

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa City Hospital, Bursa, Türkiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided